CLINICAL TRIAL: NCT00934986
Title: Study of Natural Killer Cells Function in Untreated Patients With Chronic Lymphocytic Leukemia
Brief Title: Natural Killer Cells Function in Patients With Chronic Lymphocytic Leukemia
Acronym: LLC-NK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LLC-NK/IPC 2007-004
Record Dates: First submitted 2009-07-02; First posted 2009-07-08 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; NK Cells
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Surface expression of functional biomarkers of the NK cell — An extra blood sample of 40 ml is required :
  * Stage A patient who does not require a treatment: one sample the day of enrollment.
  * Stage B or C patient who require RFC treatment: sample at D0 of the 1st and 4th cure of RFC, and 3 months after the end of the treatment.

SUMMARY:
Purpose:

The involvement of Natural Killer cells (NK) in the efficiency of the treatment in lymphoma and the beginning of new therapies based on function and activation of NK, justify an improvement of knowledge about the status of the population of NK (number, function, genic expression) in Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
Method: prospective, monocentric, descriptive study

Primary objective:

Evaluation of the expression and function of receptors activator of NK cell (KIRs) in patients with CLL at stage A with therapeutic abstention, or stage B or C which require a treatment.

Secondary objectives:

Measure of the evolution of cytotoxic function of NK cells and theirs biomarkers of activation when the patient receives an immunochemotherapy with Rituximab/ Fludarabine/ Cyclophosphamide (RCF).

Verification, by analysis, of functions and biomarkers of the adaptive and innate immunity

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL (Score of Matutes >=4) with no history of treatment: Stade A of Binet, Or Stade B or C before the beginning of the treatment with RFC
* Patients who can undergo blood collection
* Patient aged 18 years and older
* Signed consent

Non inclusion Criteria:

* Patient with anemia: haemoglobin < 9 g/dl
* Pregnancy, breast feeding
* Patient in an urgent situation, or unable to give a consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Analysis of the surface expression of functional biomarkers of the NK cell, functional study, analysis of expression of transcription of values genes. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse AURRAN-SCHLEINITZ, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut PAOLI-CALMETTES, Marseille, France

REFERENCES:
- See also: Official web site of the sponsor — http://www.institutpaolicalmettes.fr